CLINICAL TRIAL: NCT00904605
Title: A Randomized, Open-Label Study Comparing the Efficacy and Safety of Lidocaine Patch 5% With Celecoxib 200 mg in Patients With Pain From Osteoarthritis of the Knee
Brief Title: Lidocaine Patch Versus Celecoxib in Pain From Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Safety concerns with the COX-2 specific inhibitor class of drug.
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3220-012
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Lidoderm; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- Lidoderm® (Experimental): Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc.), 1⅓ patches applied topically to each affected knee every 24 hours (q24h)
  Interventions: Drug: Lidoderm
- 2-Celecoxib 200mg (Active Comparator): Celecoxib (Celebrex®, G.D. Searle & Co., Chicago, IL), one 200 mg oral capsule QD
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Lidoderm — Eligible patients were randomly allocated to receive one of two treatments for 12 weeks: lidocaine patch 5% or celecoxib 200 mg daily. Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc.), 1⅓ patches applied topically to each affected knee every 24 hours (q24h
  Arms: 1- Lidoderm®
Drug: Celecoxib — Eligible patients were randomly allocated to receive one of two treatments for 12 weeks: lidocaine patch 5% or celecoxib 200 mg daily. Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc.), 1⅓ patches applied topically to each affected knee every 24 hours (q24h)
  Arms: 2-Celecoxib 200mg

SUMMARY:
Patients with unilateral or bilateral osteoarthritis of the knee participated in a Phase IV clinical trial to assess the efficacy of Lidoderm compared with celecoxib 200mg in treating pain from osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Had unilateral or bilateral OA of the knee diagnosed according to the American College of Rheumatology (ACR) criteria based on clinical and radiographic evidence of OA (presence of osteophytes on x-ray and written evaluation)
2. Had functional capacity class rating of I, II, or III according to ACR classification
3. Had a normal 12-lead electrocardiogram (ECG) without any clinically significant abnormalities in heart rate, rhythm, or conduction
4. Had discontinued use of all analgesic medications (including over-the-counter [OTC] analgesics) prior to randomization (patients were allowed limited use of analgesic medications for non-study pain)
5. At baseline visit, patients were randomized to active treatment if they had an average daily pain intensity score for the index joint of 5 or greater (on a 0 to 10 scale) for at least 3 days out of the 5 consecutive days immediately preceding the baseline visit; 0 is defined as "no pain" and 10 is defined as "pain as bad as ever imagined" as measured by Question 5 of the BPI and recorded in a diary.
6. At baseline visit, patients were randomized to active treatment if they had an OA severity score for the index joint of 7 or greater on a composite scale of 0 to 24 as measured by the Index of Severity for Osteoarthrosis of the Knee

Exclusion Criteria:

1. Had been diagnosed with inflammatory arthritis, gout, pseudo-gout or Paget's disease that in the investigator's opinion would interfere with the assessment of pain and other symptoms of OA
2. Had elective surgery scheduled to occur during the 14-week study
3. Had serious medical conditions requiring daily medications, such as anticonvulsants and tricyclic antidepressants, that may confound study results
4. Had any other clinically significant joint disease or prior joint replacement surgery at the index joint
5. Had severe renal insufficiency (creatinine clearance of <30 mL/min)
6. Had moderate or greater hepatic impairment
7. Had experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs
8. Had a prior history of peptic ulcer disease and/or gastrointestinal bleeding
9. Were taking analgesic medications, glucosamine, or chondroitin that could not be discontinued during the study. Patients taking these medications prior to the study were required to discontinue use for the duration of the study. Patients using opioid analgesics at study entry were required to taper off these medications.
10. Were taking long-acting opioids or opioids that could not be discontinued over the first 5 days of the washout period.
11. Were receiving fluconazole or lithium (secondary to drug-drug-interaction risks)
12. Were taking a lidocaine-containing products that could not be discontinued during the study
13. Had previously failed treatment with Lidoderm analgesic patch for OA
14. Had recently received either a corticosteroid injection (within 8 weeks) or hyaluronic acid (within 6 months) of study entry
15. Were unable to discontinue use of topic drugs applied to the knee
16. Had previously failed treatment with celecoxib or with two COX-2 specific inhibitors other than celecoxib
17. Were taking class I anti-arrhythmic drugs (e.g. mexiletine, tocainide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to Week 12 in Western Ontario and McMaster Universities OA Index (WOMAC) pain subscale | Visits - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)

SECONDARY OUTCOMES:
Safety assessments included AEs, Dermal assessment (lidocaine group only), skin sensory testing (lidocaine group only), clinical laboratory test results (including urinalysis), vital sign measurements, physical examination results, body weight, plasma

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Study Director — Endo Pharmaceuticals
Locations (20):
- United States (20):
  - Hueytown, Alabama
  - Mesa, Arizona
  - Oro Valley, Arizona
  - Phoenix, Arizona
  - Carlsbad, California
  - Daytona Beach, Florida
  - Gainesville, Florida
  - Inverness, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - Decatur, Georgia
  - Marietta, Georgia
  - New Orleans, Louisiana
  - Bingham Farms, Michigan
  - Clemmons, North Carolina
  - Winston-Salem, North Carolina
  - Duncansville, Pennsylvania
  - Johnstown, Pennsylvania